CLINICAL TRIAL: NCT03077438
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Administered in Healthy Children 2 to 9 Years of Age
Brief Title: Study of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Administered in Children Aged 2 to 9 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET35; U1111 1161 2625 (Other: WHO)
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; MenACYW Conjugate vaccine; MENVEO®
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal-vaccine naïve participants aged 2 to 9 years received a single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate
- Group 2: MENVEO® Vaccine (Active Comparator): Healthy, meningococcal-vaccine naïve participants aged 2 to 9 years received a single dose of MENVEO® Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate — 0.5 milliliter (mL), Intramuscular
  Other Names: MenACYW Conjugate vaccine
  Arms: Group 1: MenACYW Conjugate Vaccine
Biological: Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: MENVEO®
  Arms: Group 2: MENVEO® Vaccine

SUMMARY:
The purpose of the study was to evaluate the immunogenicity and describe the safety of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine compared to the licensed Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 (MENVEO®) vaccine in children 2 to 9 years of age in the United States (US) and Puerto Rico.

Primary objective:

- To demonstrate the non-inferiority of the vaccine seroresponse to meningococcal serogroups A, C, Y, and W following the administration of a single dose of MenACYW Conjugate vaccine compared to that observed following the administration of a single dose of MENVEO® in children aged 2 to 9 years.

Secondary objectives:

* To compare the serum bactericidal assay using human complement (hSBA) antibody geometric mean titers (GMTs) of meningococcal serogroups A, C, Y, and W following the administration of MenACYW Conjugate vaccine to those observed following the administration of MENVEO® in children 2 to 9 years of age.
* To evaluate the hSBA antibody GMTs of meningococcal serogroups A, C, Y, and W following the administration of MenACYW Conjugate vaccine and those observed following the administration of MENVEO® in children 2 to 5 years of age, and in children 6 to 9 years of age, respectively.
* To evaluate the hSBA vaccine seroresponse to meningococcal serogroups A, C, Y, and W before and 30 days (+14 days) post-vaccination in children 2 to 5 years of age, and in children 6 to 9 years of age, respectively.

Observational objective:

- To describe the safety profile of MenACYW Conjugate vaccine and that of the licensed MENVEO®.

DETAILED DESCRIPTION:
Healthy children were randomized and received a single dose of either MenACYW Conjugate vaccine or MENVEO®. They were assessed for immunogenicity at baseline (pre-vaccination) and at 30-44 days post-vaccination. Safety information were collected post-vaccination and throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 9 years on the day of inclusion.
* Assent form had been signed and dated by the participant (as required by local regulations) and informed consent form had been signed and dated by parent(s) or guardian.
* Participant and parent/guardian were able to attend all scheduled visits and complied with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche.
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which might be received at least 2 weeks before or after the study investigational vaccines. This exception included monovalent, multivalent, live, and attenuated influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (ie., mono- or polyvalent, polysaccharide, or Conjugate meningococcal vaccine containing serogroups A, C, Y, W; or meningococcal B serogroup containing vaccine).
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Verbal report of thrombocytopenia, contraindicating intramuscular vaccination by the Investigator's judgment.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion.
* Personal history of Guillain-Barré syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator's judgment) on the day of vaccination or febrile illness (temperature ≥100.4°F). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Officer, MD, Study Director — Sanofi Pasteur Inc.
Locations (35):
- United States (34):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Dothan, Alabama
  - Investigational Site, Tucson, Arizona
  - Investigational Site, Jonesboro, Arkansas
  - Investigational Site, Anaheim, California
  - Investigational Site, Downey, California
  - Investigational Site, Paramount, California
  - Investigational Site, San Diego, California
  - Investigational Site, Council Bluffs, Iowa
  - Investigational Site, Bardstown, Kentucky
  - Investigational Site, Nicholasville, Kentucky
  - Investigational Site, Metairie, Louisiana
  - Investigational Site, Woburn, Massachusetts
  - Investigational Site, Bridgeton, Missouri
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, Omaha, Nebraska
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Dayton, Ohio
  - Investigational Site, Fairfield, Ohio
  - Investigational Site, Grants Pass, Oregon
  - Investigational Site, Gresham, Oregon
  - Investigational Site, Erie, Pennsylvania
  - Investigational Site, Hermitage, Pennsylvania
  - Investigational Site, Goodlettsville, Tennessee
  - Investigational Site, Tullahoma, Tennessee
  - Investigational Site, Layton, Utah
  - Investigational Site, Orem, Utah
  - Investigational Site, Roy, Utah
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, South Jordan, Utah
  - Investigational Site, Syracuse, Utah
  - Investigational Site, West Jordan, Utah
  - Investigational Site, Midlothian, Virginia
- Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Baccarini CI, Simon MW, Brandon D, Christensen S, Jordanov E, Dhingra MS. Safety and Immunogenicity of a Quadrivalent Meningococcal Conjugate Vaccine in Healthy Meningococcal-Naive Children 2-9 Years of Age: A Phase III, Randomized Study. Pediatr Infect Dis J. 2020 Oct;39(10):955-960. doi: 10.1097/INF.0000000000002832. PMID 32852352
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 36 centers in the United States (US) and Puerto Rico from 17 February 2017 to 30 March 2017.
Pre-assignment Details: A total of 1000 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized in the study.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy, meningococcal-vaccine naïve participants aged 2 to 9 years received a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine on Day 0.
- Group 2: MENVEO® Vaccine: Healthy, meningococcal-vaccine naïve participants aged 2 to 9 years received a single dose of Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 (MENVEO®) Conjugate vaccine on Day 0.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Started | 499 | 501
Safety Analysis Set (SafAS) (SafAS:participants who received at least 1 dose of study vaccine(s) & had any safety data available.) | 498 | 494
Completed | 487 | 487
Not Completed | 12 | 14
Not completed — Protocol Violation | 3 | 5
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine | Total
Number analyzed (Participants) | 499 | 501 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.0 (2.33) | 6.0 (2.36) | 6.0 (2.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 236 | 481
  Male | 254 | 265 | 519
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 66 | 61 | 127
  White | 402 | 417 | 819
  More than one race | 21 | 21 | 42
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 499 | 501 | 1000

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Seroresponse Measured by Serum Bactericidal Assay Using Human Complement (hSBA) Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With Either MenACYW Conjugate Vaccine or MENVEO® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. The hSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination hSBA titers greater than or equal to (>=) 1:16 for participants with pre-vaccination hSBA titers less than (<) 1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >=1:8.
Time Frame: Day 30 (post-vaccination)
Population: Per-protocol analysis set (PPAS) defined for accessing ACYW immune response data for participants who received at least 1 dose of study vaccine and had valid post-vaccination serology result. Participants who presented pre-defined protocol deviations were excluded. Here,'Number analyzed'=participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Number analyzed (Participants) | 458 | 460
percentage of participants
  Serogroup A: number analyzed (Participants) | 455 | 458
  Serogroup A | 55.4 [50.7 to 60.0] | 47.8 [43.2 to 52.5]
  Serogroup C: number analyzed (Participants) | 458 | 458
  Serogroup C | 95.2 [92.8 to 97.0] | 47.8 [43.2 to 52.5]
  Serogroup Y: number analyzed (Participants) | 458 | 459
  Serogroup Y | 91.5 [88.5 to 93.9] | 79.3 [75.3 to 82.9]
  Serogroup W: number analyzed (Participants) | 458 | 459
  Serogroup W | 78.8 [74.8 to 82.5] | 64.1 [59.5 to 68.4]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup A; Test type: Non-Inferiority — 95% confidence interval (CI) of the difference was calculated from the Wilson Score Method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference between the 2 percentages was >-10%; Percentage Difference = 7.6, 95% CI 2-sided [1.1 to 14]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup C; Test type: Non-Inferiority — 95% CI of the difference was calculated from the Wilson Score Method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference between the 2 percentages was >-10%; Percentage Difference = 47.4, 95% CI 2-sided [42.2 to 52.2]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = 12.2, 95% CI 2-sided [7.7 to 16.7]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = 14.8, 95% CI 2-sided [8.9 to 20.5]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA Following Vaccination With Either MenACYW Conjugate Vaccine or MENVEO® Vaccine in Children 2 to 9 Years of Age
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Number analyzed (Participants) | 458 | 460
titers (1/dilution)
  Serogroup A: number analyzed (Participants) | 456 | 458
  Serogroup A | 24.8 [21.9 to 27.9] | 22.6 [19.7 to 26.0]
  Serogroup C: number analyzed (Participants) | 458 | 459
  Serogroup C | 238 [209 to 270] | 17.0 [14.3 to 20.2]
  Serogroup Y: number analyzed (Participants) | 458 | 459
  Serogroup Y | 68.8 [61.3 to 77.3] | 43.5 [37.7 to 50.4]
  Serogroup W: number analyzed (Participants) | 458 | 459
  Serogroup W | 37.5 [33.7 to 41.8] | 26.2 [23.0 to 29.9]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup A; Test type: Other; GMT Ratio = 1.09, 95% CI 2-sided [0.91 to 1.32]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup C; Test type: Other; GMT Ratio = 14, 95% CI 2-sided [11.3 to 17.3]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup Y; Test type: Other; GMT Ratio = 1.58, 95% CI 2-sided [1.31 to 1.9]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup W; Test type: Other; GMT Ratio = 1.43, 95% CI 2-sided [1.21 to 1.69]

3. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA Following Vaccination With Either MenACYW Conjugate Vaccine or MENVEO® Vaccine in Children 2 to 5 Years of Age
Description: Antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here 'Overall number of participants analyzed' = number of participants in the PPAS aged 2-5 years, and 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy, meningococcal-vaccine naïve participants aged 2 to 5 years received a single dose of MenACYW Conjugate vaccine on Day 0.
- Group 2: MENVEO® Vaccine: Healthy, meningococcal-vaccine naïve participants aged 2 to 5 years received a single dose of MENVEO® Conjugate vaccine on Day 0.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Number analyzed (Participants) | 229 | 223
titers (1/dilution)
  Serogroup A: number analyzed (Participants) | 228 | 221
  Serogroup A | 21.6 [18.2 to 25.5] | 18.9 [15.5 to 23.0]
  Serogroup C | 208 [175 to 246] | 11.9 [9.79 to 14.6]
  Serogroup Y: number analyzed (Participants) | 229 | 222
  Serogroup Y | 49.8 [43.0 to 57.6] | 36.1 [29.2 to 44.7]
  Serogroup W: number analyzed (Participants) | 229 | 222
  Serogroup W | 28.8 [24.6 to 33.7] | 20.1 [16.7 to 24.2]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup A; Test type: Other; GMT Ratio = 1.14, 95% CI 2-sided [0.883 to 1.47]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup C; Test type: Other; GMT Ratio = 17.4, 95% CI 2-sided [13.4 to 22.6]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup Y; Test type: Other; GMT Ratio = 1.38, 95% CI 2-sided [1.07 to 1.78]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup W; Test type: Other; GMT Ratio = 1.43, 95% CI 2-sided [1.12 to 1.83]

4. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA Following Vaccination With Either MenACYW Conjugate Vaccine or MENVEO® Vaccine in Children 6 to 9 Years of Age
Description: Antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here 'Overall number of participants analyzed' = number of participants in the PPAS aged 6-9 years, and 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy, meningococcal-vaccine naïve participants aged 6 to 9 years received a single dose of MenACYW Conjugate vaccine on Day 0.
- Group 2: MENVEO® Vaccine: Healthy, meningococcal-vaccine naïve participants aged 6 to 9 years received a single dose of MENVEO® Conjugate vaccine on Day 0.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Number analyzed (Participants) | 229 | 237
titers (1/dilution)
  Serogroup A: number analyzed (Participants) | 228 | 237
  Serogroup A | 28.4 [23.9 to 33.8] | 26.8 [22.0 to 32.6]
  Serogroup C: number analyzed (Participants) | 229 | 236
  Serogroup C | 272 [224 to 330] | 23.7 [18.2 to 31.0]
  Serogroup Y | 95.1 [80.2 to 113] | 51.8 [42.5 to 63.2]
  Serogroup W | 48.9 [42.5 to 56.3] | 33.6 [28.2 to 40.1]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup A; Test type: Other; GMT Ratio = 1.06, 95% CI 2-sided [0.816 to 1.38]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup C; Test type: Other; GMT Ratio = 11.5, 95% CI 2-sided [8.24 to 16]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup Y; Test type: Other; GMT Ratio = 1.84, 95% CI 2-sided [1.41 to 2.38]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup W; Test type: Other; GMT Ratio = 1.45, 95% CI 2-sided [1.16 to 1.82]

5. Secondary Outcome: Percentage of Participants Achieving Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With Either MenACYW Conjugate Vaccine or MENVEO® Vaccine in Children 2 to 5 Years of Age
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. The hSBA vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >=1:16 for participants with pre-vaccination hSBA titers <1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >=1:8.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Number analyzed (Participants) | 229 | 223
percentage of participants
  Serogroup A: number analyzed (Participants) | 227 | 221
  Serogroup A | 52.4 [45.7 to 59.1] | 44.8 [38.1 to 51.6]
  Serogroup C: number analyzed (Participants) | 229 | 222
  Serogroup C | 94.3 [90.5 to 96.9] | 43.2 [36.6 to 50.0]
  Serogroup Y: number analyzed (Participants) | 229 | 222
  Serogroup Y | 88.2 [83.3 to 92.1] | 77.0 [70.9 to 82.4]
  Serogroup W: number analyzed (Participants) | 229 | 222
  Serogroup W | 73.8 [67.6 to 79.4] | 61.3 [54.5 to 67.7]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup A; Test type: Other; Percentage Difference = 7.6, 95% CI 2-sided [-1.6 to 16.7]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup C; Test type: Other; Percentage Difference = 51.1, 95% CI 2-sided [43.5 to 57.8]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup Y; Test type: Other; Percentage Difference = 11.2, 95% CI 2-sided [4.2 to 18.1]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup W; Test type: Other; Percentage Difference = 12.5, 95% CI 2-sided [3.9 to 20.9]

6. Secondary Outcome: Percentage of Participants Achieving Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With Either MenACYW Conjugate Vaccine or MENVEO® Vaccine in Children 6 to 9 Years Age
Description: as for outcome 5
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
Number analyzed (Participants) | 229 | 237
percentage of participants
  Serogroup A: number analyzed (Participants) | 228 | 237
  Serogroup A | 58.3 [51.6 to 64.8] | 50.6 [44.1 to 57.2]
  Serogroup C: number analyzed (Participants) | 229 | 236
  Serogroup C | 96.1 [92.7 to 98.2] | 52.1 [45.5 to 58.6]
  Serogroup Y | 94.8 [91.0 to 97.3] | 81.4 [75.9 to 86.2]
  Serogroup W | 83.8 [78.4 to 88.4] | 66.7 [60.3 to 72.6]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup A; Test type: Other; Percentage Difference = 7.7, 95% CI 2-sided [-1.3 to 16.6]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup C; Test type: Other; Percentage Difference = 44, 95% CI 2-sided [36.8 to 50.6]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup Y; Test type: Other; Percentage Difference = 13.3, 95% CI 2-sided [7.6 to 19.2]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO® Vaccine; Serogroup W; Test type: Other; Percentage Difference = 17.2, 95% CI 2-sided [9.4 to 24.7]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to 30 days after vaccination. Solicited Reaction (SR) data were collected within 7 days after vaccination. Serious adverse events (SAEs) data were collected throughout the study (up to 180 days after vaccination).
Description: Analysis was performed on Safety Analysis Set. A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO® Vaccine
All-Cause Mortality (participants affected / at risk) | 0/498 | 0/494
Serious Adverse Events (participants affected / at risk) | 7/498 | 3/494
Other Adverse Events (participants affected / at risk) | 304/498 | 335/494
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=498) | Group 2: MENVEO® Vaccine (N=494)
Osteomyelitis (Infections and infestations) | 1 | 0
Partial Seizures (Nervous system disorders) | 0 | 1
Tethered Cord Syndrome (Nervous system disorders) | 1 | 0
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=498) | Group 2: MENVEO® Vaccine (N=494)
Injection Site Erythema (General disorders) | 110 | 153
Injection Site Pain (General disorders) | 188 | 206
Injection Site Swelling (General disorders) | 67 | 104
Malaise (General disorders) | 103 | 99
Pyrexia (General disorders) | 20 | 27
Pharyngitis (Infections and infestations) | 24 | 25
Pharyngitis Streptococcal (Infections and infestations) | 18 | 34
Upper Respiratory Tract Infection (Infections and infestations) | 20 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 99 | 112
Headache (Nervous system disorders) | 64 | 60
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03077438/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03077438/SAP_001.pdf